CLINICAL TRIAL: NCT03800199
Title: The Validity and Reliability of the Turkish Version of the Combined Index of Severity of Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European University of Lefke (Other)
Responsible Party: Principal Investigator, Beraat Alptug, Master Physiotherapist/ Principal Investigator, European University of Lefke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ETK00-2018-0281
Record Dates: First submitted 2019-01-07; First posted 2019-01-11 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Fibromyalgia
Keywords: health statues; observational study; questionnaire
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Questionnaire: Combined Index of Severity of Fibromyalgia (ICAF)
  Intervention: Perceptive rehabilitation
  Procedure: Assessment of reliability, acceptability, validity and responsiveness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perceptive Rehabilitation (PR-group) (Experimental): Perceptive rehabilitation group will receive a treatment that, as described by on Paolucci et al. (2015). This treatment will include small latex cones with different resistance. In each session there will be over 100 cones will be placed on a rigid wood with using elastic strips. The patient will be asked to lie down supine on the material. Patients weigh will create pressure and reaction force to his/her body. Treatments will be 2 times a week till 8 weeks. There will be in total 16 sessions.
  Interventions: Other: Perceptive rehabilitation

INTERVENTIONS:
Other: Perceptive rehabilitation — The first session will be an education session. Spinous processes will be reference line of the body and patient will lie down on cones. The therapist will ask the patient first to breathe normally and feel the pressure. This will lead the patient to relax and understand cones. Then, the patient will start with the diagrammatic breathing. After breath exercises patient will perform active exercises (include stretching, warming up and cooling down) on supervision. Exercises will include the whole body. Additional to this during the session therapist will ask about the pressure of cones and she will correct the patients' posture. At the end of all the session, the therapist will take a photo of the patients back with the aim of to document the pressure and hyperaemic areas.

SUMMARY:
The aim of the investigator's study is to determine the validity and reliability of the Turkish version of the Combined Index of Severity (ICAF) in Turkish patients with Fibromyalgia Syndrome (FMS).

DETAILED DESCRIPTION:
The original form of the Combined Index of Severity of Fibromyalgia (ICAF) will be translated into Turkish by two Turkish mother tongue translators who also speak English in advanced level. Then these translations will be combined into one translation and translated back to English. These translations will send to 7 different health professions who had experience working with FMS patients. The pre-final version will be composed and tested on a group of patients with FMS. If necessary, readjustments will be made, and the final version will be investigated in FMS patients. Acceptability was assessed in terms of refusal rate, rates of missing responses, and administration time. Reliability was assessed using Cronbach's alpha and test-retest assessments. Re-test assessments will be conducted after one week from first assessment. Content validity was assessed by examining the floor and ceiling effects and skew of the distributions. Convergent and divergent validity was assessed by examining the Pearson's correlation coefficients. In addition, the confirmatory factor analysis will be done to evaluate the validity of ICAF. Responsiveness was determined by examining effect size (ES), standardized response means (SRM) and P values generated using Wilcoxon's test.

ELIGIBILITY:
Inclusion Criteria:

* Having a Fibromyalgia diagnosis according to Wolfe et al. (2016) criteria.
* Feeling Fibromyalgia symptoms last 3 mounts

Exclusion Criteria:

* Having physical and functional problems with FMS
* Having a diagnosis of chronic pain other than FMS,
* Using medicine other than simple analgesics,
* History of cardiovascular or pulmonary diseases
* Can not read and write in Turkish language

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-04-13 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Combined Index of Severity of Fibromyalgia | Changes from baseline severity at 12 weeks.
  Composed of 59 items, measures the combined severity index of fibromyalgia divided into 4 factors: physical, emotional, social and active and passive coping.The ICAF score ranges from 0 to 84, with higher values indicating higher severity.

OTHER OUTCOMES:
Revised-Fibromyalgia Impact Questionnaire (FIQR) | Changes from baseline at 12 weeks.
  The Turkish version of FIQR will be used in this study. This questionnaire has 21 individual questions. All these questions should be answered according to the past 7 days. FIQR has divided into three sections; 'function, overall impact and symptoms'. The total FIQR score will be calculated with the sum of the three domain scores. The total score will be out of 100. The higher score means a severe impact.
Socio-demographic and clinical characteristics | Changes from baseline at 12 weeks.
  Date of birth, sex, marital status, profession, education status and time of the diagnosis of FMS will be noted.
Body Mass Index (BMI) | Changes from baseline at 12 weeks.
  Weight and height will be combined to report BMI in kg/m^2.
Stanford Health Assessment Questionnaire (HAQ) | Changes from baseline at 12 weeks.
  This questionnaire will be use to asses general health of the participants.There are 20 questions in 8 sub categories of functioning (dressing, rising, eating, walking, hygiene, reach, grip, and usual activities), 1 question is about pain and 1 question is about general health. Disability index questions has four possible answers (without any difficulty: 0, with some difficulty: 1, with much difficulty: 2, unable to do: 3). Highest score represent the worsening.
Fatigue Severity Scale (FSS) | Changes from baseline at 12 weeks.
  Turkish version of Fatigue Severity Scale (FSS) will be used in this study. This scale has 9 items. Each item should be scored (strongly disagrees) 0 to 7 (strongly agrees). The minimum score=9 and maximum score possible=63. Higher score=greater fatigue severity. The average score for all 9 items constitutes the FSS score.
Short-Form 36 (SF-36) | Changes from baseline at 12 weeks.
  The quality of life questionnaire Short Form 36 (SF-36) is multidimensional, consisting of 36 items, divided into eight scales, each scale assesses a health concept, they are: limitations in physical activities because of health problems, limitations in social activities due to physical or emotional problems, limitations in daily activities due to health problems, body pain, mental health, limitations in daily activities due to emotional problems, vitality, perception of general health. All categories have their own score out of 100. Higher scores mean a better quality of life.
Pittsburgh Sleep Quality Index (PSQI) | Changes from baseline at 12 weeks.
  Turkish version of Pittsburgh Sleep Quality Index (PSQI) will be used in this study. This is a self-reported index that has 19 items with Likert and open-ended response formats. This index should be answered according to the past month. Minimum Score "0" means "good sleep" and Maximum Score "30" means "disrupted sleep".

CONTACTS AND LOCATIONS:
Overall Officials: Beraat Alptug, MSc, Principal Investigator — European University of Lefke; Emine H. Tüzün, Prof. Dr., Principal Investigator — Eastern Mediterranean University; Levent Eker, M. D., Principal Investigator — Eastern Mediterranean University; Gülbin Ergin, PhD, Principal Investigator — European University of Lefke
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

REFERENCES:
- [Background] Paolucci T, Baldari C, Di Franco M, Didona D, Reis V, Vetrano M, Iosa M, Trifoglio D, Zangrando F, Spadini E, Saraceni VM, Guidetti L. A New Rehabilitation Tool in Fibromyalgia: The Effects of Perceptive Rehabilitation on Pain and Function in a Clinical Randomized Controlled Trial. Evid Based Complement Alternat Med. 2016;2016:7574589. doi: 10.1155/2016/7574589. Epub 2016 Jan 13. PMID 26884794